CLINICAL TRIAL: NCT03424512
Title: An Open Trial of Group Metacognitive Therapy for Anxiety and Depression in Cancer Survivors
Brief Title: Group Metacognitive Therapy for Anxiety and Depression in Cancer Survivors
Acronym: GMAC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Covid-19 halted study, reorganisation of the clincial service and staff leaving posts made recruitement to a group unfeasible
Sponsor: University of Liverpool (Other)
Collaborators: University of Manchester (Other); Liverpool University Hospitals NHS Foundation Trust (Other Government)
Responsible Party: Principal Investigator, Peter Fisher, Principal Investigator, University of Liverpool
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ULiverpool
Record Dates: First submitted 2017-10-03; First posted 2018-02-07 (Actual); Last update posted 2022-08-29 (Actual); Status verified 2022-08

CONDITIONS: Cancer; Anxiety; Depression; Quality of Life
MeSH Terms: conditions — Neoplasms; Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group Metacognitive Therapy (Experimental): Group metacognitive therapy (MCT) is a brief psychological intervention designed to be delivered in small groups of 4-8 patients over a course of six, 90 minute sessions conducted on a weekly basis
  Interventions: Behavioral: Group Metacognitive Therapy

INTERVENTIONS:
Behavioral: Group Metacognitive Therapy — Group MCT is based on a manualised protocol and is structured in the following way. In session 1, idiosyncratic case formulations based on the generic metacognitive model are developed for each participant. Socialization helps patients to understand that worry/rumination and unhelpful coping strategies are maintaining emotional distress. Patients are then introduced to, and practice well established treatment techniques to modify negative beliefs about uncontrollability of rumination/worry. Later sessions address relapse prevention and involves modifying remaining use of the 'cognitive attentional syndrome', reviewing residual conviction in positive and negative beliefs and consolidating and strengthening alternative ways of responding to negative thoughts.

SUMMARY:
This study aims to test the potential of group metacognitive therapy in alleviating emotional distress in cancer survivors. The investigators aim to find out if a group based approach is acceptable to patients and feasible to deliver in a routine clinical health psychology service.

DETAILED DESCRIPTION:
Survival rates in cancer continue to improve, with over 2 million adult cancer survivors in the United Kingdom, projected to increase to 4 million by 2030. Around 25% of these survivors require treatment for clinical levels of emotional distress. Current pharmacological treatments are not very effective and are not well tolerated by patients, who prefer psychological treatments. However, meta-analyses of well-controlled studies of psychological treatments indicate that these achieve only small effect sizes. Reflecting this limited efficacy in the face of the need for psychological treatment, the National Cancer Survivorship Research Initiative highlighted development and evaluation of practically feasible interventions for depression and anxiety in cancer survivors as an urgent research priority. It is recognised that current influential psychotherapeutic approaches need to be modified to meet the specific needs associated with cancer. However modifications have been pragmatic rather than theory-driven and have not improved efficacy.

The study addresses the stages of 'development' and 'piloting and feasibility' in Medical Research Council guidance on intervention development, albeit with a relatively well-defined starting point given existing evidence for efficacy of metacognitive therapy (MCT) in other settings and promising preliminary evidence of applicability in cancer. The investigators will conduct a phase I open trial to test the potential efficacy of group MCT in cancer survivors and the hypothesised causal metacognitive mechanisms underpinning treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Cancer diagnosis at least 6 months previously
* A score of at least 15 on the Total scale score of the Hospital Anxiety and Depression Scale (HADS)
* Sufficient understanding of English to consent and engage in therapy
* Stable on, or free from, psychotropic medication
* Minimum of 18 years old

Exclusion Criteria:

* History of psychotic disorder, learning disability, or organic mental disorder
* Risk of self-harm or suicide warranting immediate intervention
* In palliative phase of treatment
* Being considered for risk-reducing or reconstructive surgery within 1 year
* Concurrent psychological intervention for emotional distress
* Cognitive impairment precluding informed consent or participation
* Undergoing acute medical treatment (e.g. chemotherapy, radiotherapy)
* Current drug/alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-12-10 (Actual); Study Completion 2018-12-10 (Actual)

PRIMARY OUTCOMES:
Hospital Anxiety Depression Scale-Total (HADS-Total) | Change in HADS total at up to 10 weeks through study completion
  Measures severity of emotional distress

SECONDARY OUTCOMES:
Cognitive Attentional Syndrome-1 (CAS-1) | Change in CAS-1 at up to 10 weeks through study completion
  Measures severity of rumination and worry
Fear of Cancer Recurrence Inventory (FCRI) | Change in FCRI at up to 10 weeks through study completion
  Measures severity of fear of cancer recurrence
Metacognition Questionnaire-30 (MCQ-30) | Change in MCQ-30 at up to 10 weeks through study completion
  Measures a range of metacognitive beliefs
Impact of Events Scale-Revised (IES-R) | Change in IES-R at up to 10 weeks through study completion
  Measures trauma related symptoms
Functional Assessment of Cancer Therapy- General (FACT-G) | Change in FACT-G at up to 10 weeks through study completion
  Measures cancer specific quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Peter Fisher, PhD, Principal Investigator — University of Liverpool
Locations (1):
- Royal Liverpool and Broadgreen NHS Trust, Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2017-07-19): https://cdn.clinicaltrials.gov/large-docs/12/NCT03424512/Prot_000.pdf
  • Informed Consent Form (2017-09-05): https://cdn.clinicaltrials.gov/large-docs/12/NCT03424512/ICF_001.pdf